CLINICAL TRIAL: NCT01367587
Title: Safety and Gastrointestinal Effects of Multiple-Dosed Intravenous Methylnaltrexone in Healthy Human Volunteers
Brief Title: Safety and Gastrointestinal Effects of Intravenous Methylnaltrexone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 253
Record Dates: First submitted 2011-06-02; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: IV Methylnaltrexone

INTERVENTIONS:
Drug: IV Methylnaltrexone

SUMMARY:
This study evaluates the safety of multiple doses of IV MNTX in normal healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Must be male or non-pregnant female volunteers
2. Must be 18 to 65 yrs of age
3. Must have no significant active disease states

Exclusion Criteria:

1. History or current evidence of disease (cardiovascular, respiratory, endocrine, renal, hepatic, hematological, or psychiatric)
2. Illicit drug users
3. Subjects who received an experimental new drug in the past 30 days
4. Subjects with any laboratory findings outside normal limits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-04; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration of IV MNTX | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.

SECONDARY OUTCOMES:
Time to Maximum Plasma Concentration of IV MNTX | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.
Clearance of IV MNTX | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.
Half-life of IV MNTX | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.
Volume of Distribution of IV MNTX | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.
Area Under the Plasma Concentration versus Time Curve (AUC) of IV MNTX | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.
Percentage of IV MNTX Excreted in Urine | 3 weeks
  To evaluate plasma pharmacokinetics of multiple-doses of intravenous methylnaltrexone in healthy human volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States